CLINICAL TRIAL: NCT01839279
Title: A Partial-Blind, Randomized, Parallel Design Study With a Nested Crossover Comparison to Define the ECG Effects of Tizanidine Compared to Placebo and the Positive Control, Moxifloxacin, in Healthy Men and Women Using a Blinded ECG Evaluator: A Thorough ECG Trial
Brief Title: A Study to Define the ECG Effects of Tizanidine Compared to Placebo and the Positive Control, Moxifloxacin, in Healthy Men and Women Using a Blinded ECG Evaluator: A Thorough ECG Trial
Acronym: TQT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ZAN-QT-1006
Record Dates: First submitted 2013-04-22; First posted 2013-04-24 (Estimated); Results first posted 2015-06-01 (Estimated); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Spasticity
MeSH Terms: conditions — Muscle Spasticity | interventions — tizanidine; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tizanidine (Experimental): Oral dose of 2 and 4 milligram (mg) tablets
  Interventions: Drug: Tizanidine
- Placebo (Placebo Comparator): Placebo followed by a single dose 400 mg moxifloxacin tablets.
  Interventions: Drug: Placebo; Drug: Moxifloxacin
- Moxifloxacin (Active Comparator): Single dose of 400 mg moxifloxacin followed by placebo.
  Interventions: Drug: Placebo; Drug: Moxifloxacin

INTERVENTIONS:
Drug: Tizanidine
  Other Names: Zanaflex
  Arms: Tizanidine
Drug: Placebo
  Arms: Moxifloxacin; Placebo
Drug: Moxifloxacin
  Arms: Moxifloxacin; Placebo

SUMMARY:
This is a single-center, partial-blind, randomized, placebo-controlled, parallel design study with a nested crossover comparison to define the ECG effects of tizanidine compared to placebo and the positive control, moxifloxacin, in healthy men and women. The study will be conducted in a Phase 1 unit with sufficient facilities to house subjects as required by the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing potential should have a negative urine pregnancy test prior to Screening and Day -2 of the trial
* All subjects of childbearing potential must practice a highly effective method of birth control excluding oral contraceptives for the duration of the trial and up to 3 months after the last dose of investigational product. Oral contraceptives are not allowed, based on the precaution listed in the Zanaflex package insert.
* Have a body mass index (BMI) ranging between 19 and 30 kg/m2
* Comprehend and be able to provide written informed consent
* Be willing and able to comply with all trial requirements

Exclusion Criteria:

* Female who is either pregnant, breastfeeding or planning to become pregnant
* History of hypersensitivity or allergic reaction to tizanidine or moxifloxacin or any of the tablet components
* Any condition possibly affecting drug absorption, metabolism or excretion including previous surgery for removal of parts of stomach, bowel, liver, gall bladder, or pancreas
* History of Long QT Syndrome or a first-generation relative with this condition
* Evidence or history of clinically significant allergies except for untreated, asymptomatic, seasonal allergies at time of dosing, hematological, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, renal, psychiatric, or neurological disease. Determination of clinical significance is to be made at the Investigator's discretion
* History or presence of any malignant or benign neoplasm considered by the investigator to be clinically significant
* History of drug or alcohol abuse or dependence within the last year
* Have an active infectious disease

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2013-04; Primary Completion 2014-02 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mathews Adera, MD, Study Director — Acorda Therapeutics
Locations (1):
- Covance- Dallas, Dallas, Texas, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Initial Placebo and Crossover to Moxifloxacin; Initial Moxifloxacin and Crossover to Placebo: Dosing of moxifloxacin will only be analyzed for cause (if the effect of moxifloxacin is not as expected).
Period: Overall Study
Arm/Group | Tizanidine | Initial Placebo and Crossover to Moxifloxacin | Initial Moxifloxacin and Crossover to Placebo
Started | 72 | 32 | 32
QT/QTc Analysis Set | 72 | 32 | 32
PK Analysis Set | 70 | 0 | 0
Moxifloxacin/Placebo Analysis Set | 0 | 31 | 30
PK/QTc Analysis Set | 70 | 0 | 0
Completed | 59 | 30 | 30
Not Completed | 13 | 2 | 2
Not completed — Adverse Event | 4 | 1 | 1
Not completed — Withdrawal by Subject | 4 | 1 | 1
Not completed — Classified as 'Other' | 5 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population
Groups:
- Total: Total of all reporting groups
Arm/Group | Tizanidine | Initial Placebo and Crossover to Moxifloxacin | Initial Moxifloxacin and Crossover to Placebo | Total
Number analyzed (Participants) | 72 | 32 | 32 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.4 (6.75) | 34.1 (7.51) | 35.3 (7.21) | 34.0 (7.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 17 | 17 | 73
  Male | 33 | 15 | 15 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 30 | 6 | 12 | 48
  Not Hispanic or Latino | 42 | 26 | 20 | 88
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: The Primary Endpoint Will be the Baseline-adjusted, Placebo-corrected Effect on QTc (ΔΔQTc) on Day 14.
Description: Change from baseline in Cardiac Repolarization (QTc Interval) at Day 14 (Tizanidine 24 mg). Moxifloxacin was not investigational drug, it was used to assess the sensitivity of the study.
Time Frame: Baseline and Day 14
Population: QT/QTc Analysis set: Received at least 1 dose of study drug (including placebo), had measurements at baseline and on-treatment with at least 1 time point post-dose with at minimum triplicate measures giving rise to a QTc value for primary correction method. Effect of moxifloxacin was as expected. Therefore, no analysis required per Medical Monitor.
Measure: Least Squares Mean (90% Confidence Interval); unit: milliseconds (msec)
Groups:
- Tizanidine 24 mg: 60 subjects Tizanidine 24 mg single dose
- Tizanidine Placebo 24 mg: 61 subjects placebo used for the analysis.
- Tizanidine 24 mg Placebo-corrected: 60 subjects Tizanidine 24 mg single dose, 61 subjects placebo used for the analysis.
Arm/Group | Tizanidine 24 mg | Tizanidine Placebo 24 mg | Tizanidine 24 mg Placebo-corrected
Number analyzed (Participants) | 60 | 61 | 121
milliseconds (msec)
  Timepoint (Hour) 0 | -4.3 [-6.3 to -2.3] | -0.5 [-2.5 to 1.4] | -3.7 [-6.6 to -0.9]
  0.5 | -2.0 [-4.0 to 0.1] | 1.2 [-0.8 to 3.2] | -3.2 [-6.0 to -0.3]
  1 | -4.0 [-6.0 to -2.0] | 2.6 [0.6 to 4.5] | -6.6 [-9.4 to -3.8]
  1.5 | -4.7 [-6.9 to -2.6] | 2.7 [0.6 to 4.8] | -7.4 [-10.5 to -4.4]
  2 | -3.6 [-5.6 to -1.6] | 2.9 [0.9 to 4.8] | -6.4 [-9.2 to -3.6]
  4 | 1.6 [-0.4 to 3.6] | 3.4 [1.4 to 5.4] | -1.8 [-4.6 to 1.0]
  8 | -2.4 [-4.1 to -0.7] | 3.1 [1.4 to 4.8] | -5.5 [-7.9 to -3.1]
  12 | -2.0 [-3.5 to -0.5] | 1.0 [-0.5 to 2.5] | -3.0 [-5.1 to -0.8]
  24 | 0.4 [-1.3 to 2.2] | 2.6 [0.9 to 4.4] | -2.2 [-4.6 to 0.2]

2. Secondary Outcome: The Baseline-adjusted, Placebo-corrected (ΔΔQTc) on QTc Method Not Selected as Primary Endpoint.
Description: Change from baseline in Cardiac Repolarization (QTc Interval) at Day 5 (Tizanidine 8 mg). Moxifloxacin was not investigational drug, it was used to assess the sensitivity of the study.
Time Frame: Baseline and Day 5
Population: as for outcome 1
Measure: Least Squares Mean (90% Confidence Interval); unit: msec
Groups:
- Tizanidine 8 mg: 70 subjects Tizanidine 8 mg single dose.
- Tizanidine Placebo 8 mg: 63 subjects placebo used for analysis.
- Tizanidine 8 mg Placebo-corrected: 70 subjects Tizanidine 8 mg single dose, 63 subjects placebo used for analysis.
Arm/Group | Tizanidine 8 mg | Tizanidine Placebo 8 mg | Tizanidine 8 mg Placebo-corrected
Number analyzed (Participants) | 70 | 63 | 133
msec
  Timepoint (Hour) 0 | -0.8 [-2.5 to 0.8] | -0.9 [-2.7 to 0.8] | 0.1 [-2.3 to 2.5]
  0.5 | -0.4 [-2.3 to 1.4] | 0.4 [-1.5 to 2.3] | -0.8 [-3.5 to 1.8]
  1 | 0.0 [-1.9 to 1.9] | 2.3 [0.3 to 4.3] | -2.3 [-5.1 to 0.4]
  1.5 | 1.1 [-0.7 to 2.9] | 1.3 [-0.6 to 3.1] | -0.1 [-2.7 to 2.4]
  2 | -0.4 [-2.0 to 1.3] | 0.4 [-1.3 to 2.1] | -0.7 [-3.1 to 1.6]
  4 | 2.6 [1.2 to 4.0] | 1.0 [-0.5 to 2.5] | 1.6 [-0.4 to 3.6]
  8 | -1.5 [-3.1 to 0.0] | 0.6 [-1.0 to 2.3] | -2.2 [-4.4 to 0.1]
  12 | -0.1 [-1.6 to 1.4] | 0.7 [-0.9 to 2.3] | -0.8 [-3.0 to 1.5]
  24 | -0.5 [-2.0 to 1.0] | 1.4 [-0.1 to 3.0] | -1.9 [-4.1 to 0.3]

3. Secondary Outcome: Assessing the Relationship Between Changes in the QTc Interval and Plasma Levels of Tizanidine Using Concentration-effect Modeling
Description: The relationship will be quantified using a linear mixed effects model with an intercept. Data from Day 5 and Day 14 were fitted into regression model to obtain a slope of change. The measure type 'Number' followed by (90% Confidence Interval) shown in results is the slope from the linear fit.
Time Frame: Day 5, Day 14
Population: Pk/QTc Analysis set will include all subjects in the QT/QTc analysis set with at least one valid PK assessment. Effect of moxifloxacin was as expected. Therefore, no analysis required per Medical Monitor.
Measure: Number (90% Confidence Interval); unit: msec per ng/mL
Arm/Group | Tizanidine
Number analyzed (Participants) | 70
msec per ng/mL | -0.1209 [-0.1894 to -0.0524]

4. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Single Doses of 8 and 24 mg Tizanidine After Reaching Steady State.
Time Frame: 0.5, 1, 1.5, 2, 4, 8, 12 & 24 hours post dose on Days 5 (8 mg) and 14 (24 mg)
Population: PK Analysis set: all subjects from Group 1 who received at least one study drug and have at least one valid PK assessment
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Day 5 (Tizanidine 8 mg) | Day 14 (Tizanidine 24 mg)
Number analyzed (Participants) | 70 | 60
ng/mL | 11.7 (43.9) | 27.4 (42.7)

5. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Single Doses of 8 and 24 mg Tizanidine After Reaching Steady State.
Time Frame: 0.5, 1, 1.5, 2, 4, 8, 12 & 24 hours post dose on Days 5 (8 mg) and 14 (24 mg)
Population: as for outcome 4
Measure: Median (Full Range); unit: hour
Arm/Group | Day 5 (Tizanidine 8 mg) | Day 14 (Tizanidine 24 mg)
Number analyzed (Participants) | 70 | 60
hour | 1.35 [0.600 to 4.10] | 2.10 [0.600 to 4.10]

6. Secondary Outcome: Area Under the Plasma Concentration-time Curve During a Dosing Interval (AUCt) of Single Doses of 8 and 24 mg Tizanidine After Reaching Steady State.
Time Frame: 0.5, 1, 1.5, 2, 4, 8, 12 & 24 hours post dose on Days 5 (8 mg) and 14 (24 mg)
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | Day 5 (Tizanidine 8 mg) | Day 14 (Tizanidine 24 mg)
Number analyzed (Participants) | 70 | 60
ng*hr/mL | 32.4 (65.1) | 115 (52.8)

ADVERSE EVENTS:
Time Frame: Up to 23 days
Groups:
- Tizanidine: Tizanidine Arm
- Initial Placebo and Crossover to Moxifloxacin: Placebo/Moxifloxacin Arm
- Initial Moxifloxacin and Crossover to Placebo: Moxifloxacin/Placebo Arm
- Placebo and Moxifloxacin Groups Combined: Combined Moxifloxacin Arm
Arm/Group | Tizanidine | Initial Placebo and Crossover to Moxifloxacin | Initial Moxifloxacin and Crossover to Placebo | Placebo and Moxifloxacin Groups Combined
Serious Adverse Events (participants affected / at risk) | 0/72 | 0/32 | 1/32 | 1/64
Other Adverse Events (participants affected / at risk) | 44/72 | 16/32 | 23/32 | 39/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tizanidine (N=72) | Initial Placebo and Crossover to Moxifloxacin (N=32) | Initial Moxifloxacin and Crossover to Placebo (N=32) | Placebo and Moxifloxacin Groups Combined (N=64)
Ectopic Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tizanidine (N=72) | Initial Placebo and Crossover to Moxifloxacin (N=32) | Initial Moxifloxacin and Crossover to Placebo (N=32) | Placebo and Moxifloxacin Groups Combined (N=64)
NERVOUS SYSTEM DISORDERS (Nervous system disorders) | 32 | 8 | 8 | 16
SOMNOLENCE (Nervous system disorders) | 20 | 4 | 4 | 8
DIZZINESS (Nervous system disorders) | 17 | 2 | 4 | 6
HEADACHE (Nervous system disorders) | 10 | 5 | 3 | 8
PARAESTHESIA (Nervous system disorders) | 7 | 0 | 1 | 1
DIZZINESS POSTURAL (Nervous system disorders) | 4 | 0 | 1 | 1
GASTROINTESTINAL DISORDERS (Gastrointestinal disorders) | 21 | 8 | 10 | 18
NAUSEA (Gastrointestinal disorders) | 9 | 4 | 5 | 9
DRY MOUTH (Gastrointestinal disorders) | 10 | 0 | 3 | 3
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS (General disorders) | 24 | 9 | 9 | 18
FATIGUE (General disorders) | 13 | 1 | 1 | 2
APPLICATION SITE PRURITUS (General disorders) | 5 | 1 | 4 | 5
APPLICATION SITE IRRITATION (General disorders) | 5 | 3 | 1 | 4
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDERS (Musculoskeletal and connective tissue disorders) | 10 | 2 | 3 | 5
BACK PAIN (Musculoskeletal and connective tissue disorders) | 4 | 2 | 1 | 3
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 4 | 0 | 1 | 1
SKIN AND SUBCUTANEOUS TISSUE DISORDERS (Skin and subcutaneous tissue disorders) | 8 | 4 | 7 | 11
RASH (Skin and subcutaneous tissue disorders) | 5 | 1 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.